CLINICAL TRIAL: NCT06803368
Title: Research on Clinical Recovery and Maintenance Strategies for Chronic Hepatitis B
Brief Title: Research on Clinical Recovery and Maintenance Strategies for CHB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Minghui Li, Head of Department, Beijing Municipal Administration of Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRWEP2024W102170101
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Chronic Hepatitis b; Hepatitis B Vaccine
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:baseline anti-HBs titer≥100 mIU/ml (No Intervention): Patients with anti-HBs titer ≥100 mIU/ml at baseline were selected as group A
- Group B:baseline anti-HBs titer<100 mIU/ml (No Intervention): Patients with anti-HBs titer<100 mIU/ml at baseline were randomly divided into group B and group C, and group B did not receive intervention
- Group C:baseline anti-HBs titer<100 mIU/ml (Experimental): Patients with anti-HBs titer<100 mIU/ml at baseline were randomly divided into group B and group C, and group C received hepatitis B vaccine injection.
  Interventions: Biological: baseline anti-HBs titer

INTERVENTIONS:
Biological: baseline anti-HBs titer — Patients with baseline anti-HBs titer<100 mIU/ml were randomly divided into two groups, group B and group C. Group B did not intervene, while group C received hepatitis B vaccine intervention and observed its indicators.
  Arms: Group C:baseline anti-HBs titer<100 mIU/ml

SUMMARY:
Collect basic information of patients before antiviral treatment and when HBsAg disappears, and divide them into three groups A, B, and C based on baseline anti HBs titers after informed consent. During the follow-up period of all patients, clinical biochemistry, virology (HBVDNA, HBVRNA), serological indicators (HBsAg, anti HBs, HBeAg, anti HBe, HBcrAg, anti HBc), AFP, Fibroscan, liver imaging examinations will be conducted every 3-6 months, and blood samples will be retained for monitoring the frequency of immune cells (pDC, Treg) and the expression of functional molecules, as well as cytokines (IFN - γ, IP-10, IL-10, and TGF - β). Observe the sustained response rate and recurrence rate of virological and serological indicators, as well as the incidence of hepatitis and liver cancer during the follow-up period.

DETAILED DESCRIPTION:
Collect basic information of patients before antiviral treatment and when HBsAg disappears, and divide them into three groups A, B, and C based on baseline anti HBs titers after informed consent. Group A has an anti HBs titer ≥ 100mIU/ml and is followed up every 3-6 months for observation. The anti HBs titers<100mIU/ml were randomly divided into two groups: Group B and Group C. Group B did not intervene and was followed up every 3-6 months for observation; In group C, 20 micrograms of recombinant hepatitis B vaccine were injected subcutaneously three times on day 0, January and March. For group C patients, the level of anti HBs was detected at the 4th month after the initial vaccination. For those who could not produce anti HBs (anti HBs<10mIU/ml), the recombinant hepatitis B vaccine was subcutaneously injected three times, 20 μ g each time, in 0 day, January and March. During the follow-up period of all patients, clinical biochemistry, virology (HBVDNA, HBVRNA), serological indicators (HBsAg, anti HBs, HBeAg, anti HBe, HBcrAg, anti HBc), AFP, Fibroscan, liver imaging examinations were conducted every 3-6 months, and blood samples were retained for monitoring the frequency of immune cells (pDC, Treg) and the expression of functional molecules, as well as cytokines (IFN - γ, IP-10, IL-10, and TGF - β). Observe the sustained response rate and recurrence rate of virological and serological indicators, as well as the incidence of hepatitis and liver cancer during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old;
* Gender is not limited;
* CHB patients who meet the diagnostic criteria of the 2019 edition of the Guidelines for the Prevention and Treatment of Chronic Hepatitis B [5];
* Confirmed interferon treatment resulted in HBsAg disappearance, HBeAg negativity, and HBV DNA below the lower detection limit and cessation Patients treated with interferon;
* Sign a written informed consent form.

Exclusion Criteria:

* Merge with other hepatitis virus (HCV, HDV) infections;
* Autoimmune liver disease;
* HIV infection;
* Long term alcohol abuse and/or other liver damaging drugs;
* Mental illness;
* Evidence of liver tumors (liver cancer or AFP>100ng/ml);
* Decompensated cirrhosis;
* Individuals with serious diseases of the heart, brain, lungs, kidneys, and other systems who cannot participate in long-term follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response rate and relapse rate by virological and serological indicators | Conduct testing every 3-6 months
  The levels of biochemical, AFP, HBV DNA, HBV RNA, HBsAg, anti-HBs, HBeAg, anti-He, anti-He, HBcrAg and anti-HBc measured the expression of frequency and functional molecules of peripheral blood pDC and Treg cells and the plasma levels of IFN- γ, IP-10, IL-10 and TGF- β

SECONDARY OUTCOMES:
The incidence of hepatitis and liver cancer | 36 months
  The incidence of hepatitis and liver cancer among the enrolled researchers during the research process
  The incidence of hepatitis and liver cancer among the enrolled researchers during the research process
  The incidence of hepatitis and liver cancer among the enrolled researchers during the research process.

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Li, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Beijing, Beijing Municipality, China